CLINICAL TRIAL: NCT03841175
Title: Forecasts Impact of the Pre-therapeutic TEP-TDM in the 18-FDG Restaging of Upper Aero-digestive Tract Cancers
Acronym: RENOVATE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RENOVATE ( 29BRC18.0012)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-04

CONDITIONS: Cancer of Head and Neck
Keywords: Squamous cell carcinoma; FDG PET/CT; Initial staging; Clinical management; Prognosis
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck (HN) cancer is the sixth most common malignancy worldwide, with around 800 000 new cases and 320 000 deaths in 2015. These malignancies encompass cancers of the oral cavity, oropharynx, hypopharynx and larynx and concern squamous cell carcinomas (HNSCC) 90% of the time. Despite aggressive treatment strategies, the five-year survival rate has only marginally improved in the past decade. The prognosis is strongly dependent on initial staging. The 5-year relative survival rate is 80,3% for patients with localized disease whereas it decreases to 47.2% when regional lymph node metastasis is known, and to 32.5% when distant metastasis is known. Hence, precise cancer staging is essential as it allows clinicians to select the appropriate treatment strategies and predict the prognosis of the patients.

The conventional work-up (CWU) includes physical examination, endoscopy, computed tomography (CT) and/or magnetic resonance imaging (MRI) of the head and neck to evaluate the initial local and regional HNSCC staging. Thoracic CT is recommended because the thorax is the most frequent location of remote metastasis and synchronous second cancer outside of the upper aerodigestive tract.

Some authors demonstrated that 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) had a higher sensitivity and specificity for determining the extent of the disease and was able to detect occult second primaries. Moreover 18-FDG PET-CT allows whole body assessment. This is why the use of 18-FDG PET-CT has increased significantly over the last several years. Added to initial CWU, 18-FDG PET-CT may restage HNSCC and as a result may alter the clinical management.

Pre-therapeutic 18F-FDG PET/CT is recommended by guidelines to assess remote extension of locally advanced HNSCC and/or to look for synchronous cancer but is not systematically indicated, particularly for localized disease.

Restaging impact on prognosis and clinical management remains poorly understood.

Therefore, the objective of this study is to assess the impact of the additional information provided by 18F-FDG PET-CT on HNSCC initial staging and whether restaging modify prognosis and clinical management, whatever the CWU stage.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven HSNCC
* written consent

Exclusion Criteria:

* previous head and neck malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred for a pre-treatment FDG PET/CT of biopsy proven HSNCC
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Prognostic impact of initial restaging HNSCC with 18F-FDG PET-CT | 10 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France